CLINICAL TRIAL: NCT02383758
Title: An Interdisciplinary Approach to the Treatment of Encopresis in Children With Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Organization for Autism Research (Other)
Responsible Party: Principal Investigator, Nathan A. Call, Ph.D., BCBA-D, Instructor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00076608
Record Dates: First submitted 2015-02-25; First posted 2015-03-09 (Estimated); Results first posted 2018-01-11 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-05

CONDITIONS: Encopresis; Autistic Disorder
Keywords: Behavioral Symptoms; Child Development Disorders, Pervasive; Bowel Incontinence; Constipation
MeSH Terms: conditions — Encopresis; Autistic Disorder; Behavioral Symptoms; Child Development Disorders, Pervasive; Fecal Incontinence; Constipation | interventions — Sennosides

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Program (Experimental): Pediatric subjects with autistic spectrum disorder will begin treatment immediately. The treatment program will consist of 10 appointments of up to 4 hours each, over a 14 day period, followed by 4 weekly 1-hour follow-up visits. During each appointment, subjects will be guided to sit on the toilet. If the participant has a continent urination they will be provided with praise and remain on the toilet. If a participant has a continent bowel movement they will be provided with enthusiastic praise along with positive reinforcement and they will be allowed to leave the bathroom. A continent bowel movement will end that day's appointment. If necessary, glycerin suppositories, bisacodyl suppositories, and/or senna may be used to aid in the bowl movement.
  Interventions: Drug: Glycerin Suppository; Drug: Bisacodyl suppository; Drug: Senna
- Waitlist Control (Active Comparator): Pediatric subjects with autistic spectrum disorder will wait for 8 weeks and then be offered treatment at that time.The treatment program will consist of 10 appointments of up to 4 hours each, over a 14 day period, followed by 4 weekly 1-hour follow-up visits. During each appointment, participants will be guided to sit on the toilet. If the participant has a continent urination they will be provided with praise and remain on the toilet. If a participant has a continent bowel movement they will be provided with enthusiastic praise along with positive reinforcement and they will be allowed to leave the bathroom. A continent bowel movement will end that day's appointment. If necessary, glycerin suppositories, bisacodyl suppositories, and/or senna may be used to aid in the bowl movement.
  Interventions: Drug: Glycerin Suppository; Drug: Bisacodyl suppository; Drug: Senna

INTERVENTIONS:
Drug: Glycerin Suppository — Nursing staff will administer one glycerin suppository in the bathroom if there is no continent bowl movement in the first 30 minutes. Subjects will be taken to the bathroom 5 minutes after the suppository is administered for a 30 minute sit or until a continent void occurs. If continent bowel movements maintain on two subsequent days (after bisacodyl suppositories are discontinued) the glycerin suppository will be discontinued. At least one primary caregiver will be trained on all components of intervention still in use on the last day their child's admission. Four weekly follow-up appointments will be used to support them as they continue to implement the protocol at home, including continuing to fade out the use of medications for participants who are at least partially continent but not fully independent at the time of discharge.
Drug: Bisacodyl suppository — If a subject does not have a bowel movement during the 30 minute sit following administration of the glycerin suppository, they will be given a 1 hour break, after which a bisacodyl suppository will be administered. The participant will then sit for an additional 30 minutes.If continent bowel movements maintain for two subsequent days (after senna is discontinued) bisacodyl suppositories will be discontinued if it was required. At least one primary caregiver will be trained on all components of intervention still in use on the last day their child's admission. Four weekly follow-up appointments will be used to support them as they continue to implement the protocol at home, including continuing to fade out the use of medications for participants who are at least partially continent but not fully independent at the time of discharge.
Drug: Senna — If no continent bowel movements occur for two consecutive treatment days, caregivers will be asked to administer senna each evening thereafter until medication tapering begins. Once there have been two successive days with continent bowel movements, senna will be removed from the intervention if it was required.

SUMMARY:
The purpose of this study is to try to treat bowel movement (BM) accidents differently with children with autism spectrum disorder (ASD). The study will use over-the-counter (OTC) medications to evoke predictable bowel movements. This will make it possible for investigators to use certain strategies to reward BMs in the toilet. Independence will be increased by fading out the use of medications. The investigators will also train caregivers to implement the procedures.

DETAILED DESCRIPTION:
A large percentage of individuals with autism spectrum disorder (ASD) are delayed in achieving continence with bowel movements or never achieve it at all (i.e., they meet criteria for encopresis). This problem has tremendous ramifications for these individuals and their families because encopresis restricts them from integration with peers, limits access to educational opportunities, and carries significant social stigma. Previous interventions for encopresis in this population have either been unsuccessful or required implementation over very long periods.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-21
* Confirmed diagnosis of autistic spectrum disorder using the Social Communication Questionnaire (SCQ) and the Childhood Autism Rating Scale II (CARSII)
* Clearance from gastroenterologist for use of glycerin suppository, bisacodyl suppository and senna
* Caregiver willing to give consent/assent

Exclusion Criteria:

* Age under 5 year or over 21 years
* Does not present a diagnosis of autistic spectrum disorder
* Previous intestinal surgeries or concurrent enuresis
* Caregiver unwilling to give consent/assent

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Call, PhD, Principal Investigator — Emory University
Locations (1):
- Marcus Autism Center, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between February 2015 and January 2017.
Pre-assignment Details: Of the 22 subjects consented for participation, 20 were randomized to a study intervention and were included in study analyses.
Groups:
- Treatment Program: Pediatric subjects with autistic spectrum disorder were randomized to participate in the encopresis treatment program immediately.
  Glycerin Suppository: Nursing staff administered one glycerin suppository in the bathroom if there was no continent bowl movement in the first 30 minutes.
  Bisacodyl suppository: If a subject did not have a bowel movement during the 30 minute sit following administration of the glycerin suppository, they were given a 1 hour break, after which a bisacodyl suppository was administered.
  Senna: If no continent bowel movements occurred for two consecutive treatment days, caregivers were asked to administer senna each evening thereafter until medication tapering began.
- Waitlist Control: Pediatric subjects with autistic spectrum disorder were randomized to participate in the encopresis treatment program 8 weeks after providing consent.
  Glycerin Suppository: Nursing staff administered one glycerin suppository in the bathroom if there was no continent bowl movement in the first 30 minutes.
  Bisacodyl suppository: If a subject did not have a bowel movement during the 30 minute sit following administration of the glycerin suppository, they were given a 1 hour break, after which a bisacodyl suppository was administered.
  Senna: If no continent bowel movements occurred for two consecutive treatment days, caregivers were asked to administer senna each evening thereafter until medication tapering began.
Period: Overall Study
Arm/Group | Treatment Program | Waitlist Control
Started | 10 | 10
Completed | 10 | 8
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Participants randomized to an intervention arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Program | Waitlist Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 10 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 10 | 6 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percent Continent
Description: The percentage of participant's with continent bowel movements (control of passage of stool from the bowel).
Time Frame: Baseline, Post-Intervention (Week 2) , Follow Up (Week 4)
Population: An intention to treat (ITT) analysis was conducted; all participants who were enrolled and randomly allocated to treatment are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Program | Waitlist Control
Number analyzed (Participants) | 10 | 10
percentage of participants
  Baseline | 0 | 0
  Post-Intervention (Week 2) | 6 | 0
  Follow Up (Week 4) | 5 | 0

2. Secondary Outcome: Percent Independence
Description: Percent independence is the percentage of independent bowel movements recorded by a caregiver. A continent bowel movement without the use of any medications will constitute an independent bowel movement.
Time Frame: Baseline, Post-Intervention (Week 2) , Follow Up (Week 4)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Program | Waitlist Control
Number analyzed (Participants) | 10 | 10
percentage of participants
  Baseline | 0 | 0
  Post-Intervention (Week 2) | 0 | 0
  Follow Up (week 4) | 5 | 0

3. Secondary Outcome: Mean Clinical Global Impression for Severity (CGI-S) Score
Description: An independent evaluator (IE) will use the parent target problem (PTP) interview to help caregivers estimate the frequency of encopresis as well as its impact on the family. From this description, the IE (who will be blind to treatment assignment) will generate a brief narrative describing the participant's encopresis. This narrative will be used by the IE to rate the overall severity on the 7-point Clinical Global Impression for Severity (CGI-S). Clinical Global Impression of Severity (CGI-S) Scale is a clinician's assessment of patient's severity of illness. The score ranges from 1 = normal, not at all ill to 7 = among the most extremely ill patients
Time Frame: Baseline, Post-Intervention (Week 6), Post-Intervention (Week 10)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Program | Waitlist Control
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline | 5.4 (.7) | 5.2 (.4)
  Post-Intervention (Week 6) | 5.0 (.9) | 5.0 (.5)
  Post-Intervention (Week 10) | 4.3 (.9) | 4.9 (.6)

4. Secondary Outcome: Mean Clinical Global Impression for Improvement (CGI-I) Score
Description: An independent evaluator (IE) will use the parent target problem (PTP) interview to help caregivers estimate the frequency of encopresis as well as its impact on the family. From this description, the IE (who will be blind to treatment assignment) will generate a brief narrative describing the participant's encopresis. This narrative will be used by the IE to rate the overall severity on the 7-point Clinical Global Impression for Improvement (CGI-I). Clinical Global Impression for Improvement (CGI-I) Scale is a clinician's assessment of a patient's change in condition from baseline.The score ranges from 0 = not assessed, 1 = very much improved, through 7 = very much worse.
Time Frame: Post-Intervention (Week 6), Post-Intervention (Week 10)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Program | Waitlist Control
Number analyzed (Participants) | 10 | 10
units on a scale
  Post-Intervention (Week 6) | 3.0 (.5) | 3.8 (.6)
  Post-Intervention (Week 10) | 2.1 (.9) | 3.6 (1.0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the duration of the study (1 year and 11 months).
Arm/Group | Treatment Program | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
This is a pilot trial with a limited sample size. Outcome measure percent change in the number of bowel movements/day was adjusted due to percentage of patients continent due to most participants having no bowel movements at baseline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes